CLINICAL TRIAL: NCT03328104
Title: Aflac LL1602 ENCERT: A Phase 1 Trial Using Everolimus in Combination With Nelarabine, Cyclophosphamide and Etoposide in Relapsed T Cell Lymphoblastic Leukemia/Lymphoma
Brief Title: Everolimus in Combination With Nelarabine, Cyclophosphamide and Etoposide in Lymphoblastic Leukemia/Lymphoma
Acronym: ENCERT
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Himalee Sabnis, Assistant Professor, Emory University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: IRB00095500
Record Dates: First submitted 2017-10-20; First posted 2017-11-01 (Actual); Last update posted 2023-07-21 (Actual); Status verified 2023-07

CONDITIONS: Lymphoblastic Leukemia; Lymphoblastic Lymphoma
Keywords: T- cell acute lymphoblastic leukemia; T-ALL; T-cell lymphoblastic lymphoma; T-LLy; Everolimus; Maximum tolerated dose
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma; Precursor T-Cell Lymphoblastic Leukemia-Lymphoma | interventions — Everolimus; nelarabine; Cyclophosphamide; Etoposide

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Everolimus in combination with standard chemotherapy (Experimental): A treatment course lasts 28 days, during which participants take everolimus by mouth every day and also get standard chemotherapy via IV on certain days.
  Interventions: Drug: Everolimus; Drug: Nelarabine; Drug: Cyclophosphamide; Drug: Etoposide

INTERVENTIONS:
Drug: Everolimus — Given once daily orally via mouth or NG tube beginning at Dose Level (DL) 1 (4 mg/m2/day). Depending on safety and tolerability, dose levels will be escalated to DL2 (5 mg/m2/day). There is also a dose level de-escalation to DL0 (3 mg/m2/day) if toxicity is noted at DL1. Begins at Day 1 through 28.
Drug: Nelarabine — 650 mg/m2 IV daily x Day 1-5
Drug: Cyclophosphamide — 440 mg/m2 IV x Day 1-5
Drug: Etoposide — 100 mg/m2 IV x Day 1-5

SUMMARY:
T- cell acute lymphoblastic leukemia (T-ALL) or T-cell lymphoblastic lymphoma (T-LLy) has an increase in proteins in a specific pathway called the mTOR pathway within the cancer cells. In cancer cells it can encourage untimely cell growth, cell production, and cell survival. Everolimus is an inhibitor of the mTOR pathway and can decrease the growth and survival of cancer cells. It also prevents communication within cells and stops proteins from being made that may contribute to leukemia. The main purpose of the study is to find the maximum tolerated dose of everolimus when used together with standard chemotherapy.

DETAILED DESCRIPTION:
T- cell acute lymphoblastic leukemia (T-ALL) or T-cell lymphoblastic lymphoma (T-LLy) has an increase in proteins in a specific pathway called the mTOR pathway within the cancer cells. In cancer cells it can encourage untimely cell growth, cell production, and cell survival. Everolimus is an inhibitor of the mTOR pathway and can decrease the growth and survival of cancer cells. It also prevents communication within cells and stops proteins from being made that may contribute to leukemia.

Two to six participants will receive the starting dose of everolimus. If the side effects are not too severe, the next group of participants will take the study drug at a higher dose level. Up to two dose levels of the study drug will be tested. The main purpose of the study is to find the maximum tolerated dose of everolimus when used together with standard chemotherapy. Everolimus has been found to be safe and effective in adults and children for treatment of T- and B-cell leukemias and lymphomas.

ELIGIBILITY:
Inclusion Criteria:

1.1 Age: Subjects must be > than 1 year and < 30 years of age at the time of study enrollment.

1.2 Diagnosis Leukemia

Patients must have relapsed (first or greater relapse) or refractory T-cell acute lymphoblastic leukemia (T-ALL) with:

1. Relapsed T-ALL with an M2 (blasts ≥ 5 to ≤ 25%) or M3 (>25% blasts) marrow with or without an extramedullary site of relapse; including CNS 2 OR
2. Refractory disease after induction failure of newly diagnosed patients OR no more than two more cycles of therapy OR
3. Refractory disease with no more than one prior salvage attempt following the current relapse

Lymphoma

Patients must have relapsed (first or greater relapse) or refractory lymphoma with:

1. Lymphoblastic lymphoma or peripheral T-cell lymphoma.
2. Histologic verification of disease at original diagnosis or subsequent relapse.
3. Evaluable or measurable disease documented by clinical or radiographic criteria or bone marrow disease present at study entry.
4. Patient may have CNS 2 status if other sites of leukemia or lymphoma involvement are present.

   1.3 Performance Score Patients must have a Karnofsky ≥ 50% for subjects > 16 years of age and Lansky score ≥ 50 for subjects ≤ 16 years of age (See Appendix I).

   Note: Subjects who are unable to walk because of paralysis, but who are up in a wheelchair, will be considered ambulatory for the purpose of assessing the performance score.

   1.4 Prior Therapy A. Patients who relapse while receiving standard ALL maintenance chemotherapy will not be required to have a waiting period before entry onto this study.

   B. Patients who relapse on therapy other than standard ALL maintenance therapy must have fully recovered from the acute toxic effects of all prior chemotherapy, immunotherapy, or radiotherapy prior to entering this study.
   * Cytotoxic Chemotherapy: At least 7 days must have elapsed since the completion of cytotoxic therapy (other than standard ALL maintenance therapy as per 4.1.4.B) with the exception of hydroxyurea, which is permitted up to 24 hours prior to the start of protocol therapy.
   * Nitrosureas: At least 42 days must have elapsed since administration of nitrosureas.
   * Hematopoietic growth factors: At least 14 days after the last dose of long acting hematopoietic growth factor (e.g. Neulasta) or 7 days for short acting growth factor (e.g. Neupogen)
   * Radiation: At least 84 days must have elapsed since administration of craniospinal, hemipelvic or other radiation therapy to more than 25% of the bone marrow containing spaces. At least 42 days must have elapsed if other substantial marrow radiation has been given.
   * Nelarabine Prior therapy: Patients who have previously been treated with nelarabine are eligible, however if they have previously received a regimen of nelarabine, cyclophosphamide and etoposide, they are not eligible.
   * Biologic (anti-neoplastic agent): At least 7 days after the last dose of a biologic agent. For agents that have known adverse events occurring beyond 7 days after administration, this period must be extended beyond the time during which adverse events are known to occur. The duration of this interval must be discussed with the study chair
   * Immunotherapy: At least 42 days after the completion of any type of immunotherapy (e.g., tumor vaccines or chimeric antigen receptor T cell (CART) therapy
   * Monoclonal Antibodies: Monoclonal antibodies: At least 3 half-lives of the antibody must have elapsed after the last dose of a monoclonal antibody (See Appendix II for details)
   * Stem Cell Infusion: No evidence of active graft vs. host disease and at least 84 days must have elapsed after transplant or stem cell infusion.
   * Study specific limitations on prior therapy: Patient may not have previously received therapy with an mTOR inhibitor.
   * Prior Intrathecal Therapy: Patients may be enrolled on study regardless of the timing of prior Intrathecal therapy; however, they MAY NOT BEGIN TREATMENT ON THIS PROTOCOL UNTIL A MINIMUM OF 7 DAYS HAS ELAPSED SINCE PRIOR INTRATHECAL THERAPY.

   1.5 Adequate organ function

   A. Adequate Bone Marrow Function Defined as:

   • Patients should not be known to be refractory to red blood cell or platelet transfusions.

   • Blood counts are not required to be normal prior to enrollment on trial.

   B. Adequate Hepatic Function defined as:

   • Total bilirubin (sum of conjugated + unconjugated) ≤ 1.5 x institutional upper limit of normal for age
   * SGPT (ALT) and SGOT (AST) must be ≤ 3 x institutional upper limit of normal (Grade 1 or less per CTCAE 4).
   * GGT must be ≤ 2.5 x institutional upper limit of normal (Grade 1 or less per CTCAE 4).
   * Serum albumin ≥ 2 g/dL.
   * The hepatic requirements may be waived for patients with Grade 1 or 2 elevations of hepatic transaminases clearly due to leukemic infiltration after consultation with a study Co-Chair.

   C. Adequate Renal Function defined as:

   • Serum creatinine ≤ 1.5x upper limit of normal (ULN) for age. If the serum creatinine is above these values, the calculated creatinine clearance or radioisotope GFR must be ≥ 70 mL/min/1.73m2.

   D. Adequate Cardiac Function defined as:
   * Shortening fraction of ≥ 27% by echocardiogram, OR
   * Ejection fraction of ≥ 50% by gated radionuclide study/echocardiogram

   E. Adequate Pulmonary Function defined as:
   * Pulse oximetry > 94% on room air
   * No evidence of dyspnea at rest and no exercise intolerance.
   * Baseline chest x-ray with no evidence of active infectious disease or pneumonitis.

   F. Reproductive Function

   • Female patients of childbearing potential must have a negative urine or serum pregnancy test confirmed prior to enrollment.
   * Female patients with infants must agree not to breastfeed their infants while on the study.
   * Male and female patients of child-bearing potential must agree to use an effective method of contraception approved by the investigator during the study.

   G. Normal blood glucose levels as defined as:
   * Fasting or random blood glucose within the upper limits of normal for age.
   * If random blood glucose is above upper limits for age, a fasting blood glucose can be obtained and must be within normal limits for age

   H. Normal triglyceride and cholesterol as defined as:

   • Fasting or non-fasting serum triglyceride level ≤ 300 mg/dL and serum cholesterol level ≤ 300 mg/dL.

   1.6 Informed Consent Patients and/or their parents or legal guardians must be capable of understanding the investigational nature, potential risks and benefits of the study. All patients and/or their parents or legal guardians must sign a written informed consent. Age appropriate assent will be obtained per institutional guidelines. To allow non-native speaking patients to participate in this study, bilingual health services will be provided in the appropriate language, when feasible, according to individual institutional practices and guidelines

   1.7 Protocol Approval All institutional, local, state, FDA, and OHRP requirements for human studies must be met.

   Exclusion Criteria:

   2.1 Diagnosis

   • Patients with CNS3 disease as defined in section 4.3.1

   • Patients with isolated extra-medullary relapse involving only sanctuary sites (eg. Testicular relapse) but patients with extramedullary disease involving nodal or other non-sanctuary sites are eligible

   • Patients with isolated testicular relapse

   • Patients with Ph+ T-ALL/T-LLy
   * Patients with Down Syndrome
   * Patients with pre-existing Grade 2 (or higher) peripheral motor or sensory neurotoxicity per CTCAE 4.03
   * Patients with a history of prior veno-occlusive disease (VOD)/sinusoidal obstruction syndrome (SOS) or findings consistent with a diagnosis of VOD/SOS, defined as: conjugated serum bilirubin >1.4 mg/dL AND unexplained weight gain greater than 10% of baseline weight or ascites AND hepatomegaly or right upper quadrant pain without another explanation, OR reversal of portal vein flow on ultrasound, OR pathological confirmation of VOD on liver biopsy.

   2.2 Infection Criteria

   • Positive blood culture within 48 hours of study enrollment;

   • Fever above 38.2 within 48 hours of study enrollment with clinical signs of infection. Fever that is determined to be due to tumor burden is allowed if patients have documented negative blood cultures for at least 48 hours prior to enrollment and no concurrent signs or symptoms of active infection or hemodynamic instability.

   • Active fungal, viral, bacterial, or protozoal infection requiring IV treatment. Chronic prophylaxis therapy to prevent infections is allowed

   2.3 Skin condition Patients with pre-existing Grade 1 or higher ulcerations, fistulas, mucosal lesions, or skin barrier breakdown

   2.4 Concomitant Medications
   * Corticosteroids: Patients receiving corticosteroids who have not been on a stable or decreasing dose of corticosteroid for at least 7 days prior to enrollment are not eligible. Corticosteroids must be held for 24 hours prior to initiation of study therapy.
   * Investigational Drugs: Patients who are currently receiving another investigational drug are not eligible. The definition of "investigational" for use in this protocol means any drug that is not licensed by the FDA
   * Anti-cancer agents: Patients who are currently receiving or may receive while on therapy, other anti-cancer agents, radiation therapy or immunotherapy are not eligible [except leukemia patients who relapsed on Maintenance therapy or patients receiving hydroxyurea, which may be continued until 24 hours prior to start of protocol therapy]. Intrathecal therapy may be given up to one week prior to initiation of study treatment.
   * Anti-GVHD or agents to prevent organ rejection post-transplant: Patients who are receiving cyclosporine, tacrolimus or other agents to prevent either graft-versus-host disease post bone marrow transplant or organ rejection post-transplant are not eligible for this trial. At least 3 half-lives must have elapsed after the last dose of GVHD meds.
   * Angiotensin-converting enzyme (ACE) inhibitors: Patients who are currently receiving ACE inhibitors are not eligible due to the development of angioneurotic edema-type reactions in some subjects who received concurrent treatment with everolimus + ACE inhibitors. At least 3 half-lives must have elapsed after the last dose of ACE inhibitors.
   * Anti-convulsants: Patients who are currently receiving CYP3A4/PgP enzyme inducing anticonvulsants (eg. phenytoin, phenobarbitol, or carbamazepine) are not eligible. Stabilizing on a non-hepatic inducing metabolizing anti-convulsant (ie: gabapentin or levetiracetam) prior to study entry is acceptable. At least 3 half-lives must have elapsed after the last dose of enzyme inducing anti-convulsants.
   * Inhibitors of everolimus metabolism: Patients receiving treatment with azoles such as fluconazole or voriconazole which are potent inhibitors of everolimus metabolism. At least 3 half-lives must have elapsed after the last dose of azoles.

   2.5 Patients with significant concurrent disease, illness, psychiatric disorder or social issue that would compromise patient safety or compliance with protocol treatment or required observations, interfere with consent, study participation, follow up, or interpretation of study results.

Ages: 2 Years to 29 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 8 (Actual)
Dates: Start 2018-07-24 (Actual); Primary Completion 2023-06-29 (Actual); Study Completion 2023-06-29 (Actual)

PRIMARY OUTCOMES:
Determine the maximum tolerated dose (MTD). | Day 1-29
  Maximum Tolerated Dose (MTD) will be defined as the highest dose level tested at which 0/6 or 1/6 patients experience Dose Limiting Toxicity (DLT) with at least 2/3 or 2/6 patients encountering DLT at the next higher dose.

SECONDARY OUTCOMES:
Determine area under the concentration versus time curve (AUC) | Day 1, 8 and 15 of course 1
  Blood will be collected on day 1, 8 and 15 of course 1 to determine the levels of everolimus in the body. On each of the three days, levels will be determined 30 min prior to administration of everolimus (hr 0), and 2, 6 and 24 hours after administration of everolimus. Everolimus concentrations will be measured by liquid chromatography/mass spectrometric analysis following a high throughput liquid/liquid extraction. Professional software and standard noncompartmental methods will be used to calculate area under the concentration versus time curve (AUC).
Determine maximum observed concentration (Cmax) | Day 1, 8 and 15 of course 1
  Blood will be collected on day 1, 8 and 15 of course 1 to determine the levels of everolimus in the body. On each of the three days, levels will be determined 30 min prior to administration of everolimus (hr 0), and 2, 6 and 24 hours after administration of everolimus. Everolimus concentrations will be measured by liquid chromatography/mass spectrometric analysis following a high throughput liquid/liquid extraction. Professional software and standard noncompartmental methods will be used to calculate maximum observed concentration (Cmax).
Determine elimination half-life (t1/2) | Day 1, 8 and 15 of course 1
  Blood will be collected on day 1, 8 and 15 of course 1 to determine the levels of everolimus in the body. On each of the three days, levels will be determined 30 min prior to administration of everolimus (hr 0), and 2, 6 and 24 hours after administration of everolimus. Everolimus concentrations will be measured by liquid chromatography/mass spectrometric analysis following a high throughput liquid/liquid extraction. Professional software and standard noncompartmental methods will be used to calculate elimination half-life (t1/2).
Changes in phosphoprotein (pAkt and p4EBP1) expression at time points pre- and post everolimus therapy in peripheral blood mono-nuclear cells (PBMCs) and bone marrow. | Day 1, 8 and 15 and day 29/ at count recovery at the end of course 1 (whichever is earlier)
  Levels of phosphorylated p-Akt and p-4EBP1 will be determined in PBMC's using nano-immunoassay. Mean levels of p-Akt and p-4EBP1 will be calculated at each time point and compared with response at the end of course 1 using repeated measures ANOVA.
Changes in Mer expression at time points pre- and post everolimus therapy in peripheral blood mono-nuclear cells (PBMCs) and bone marrow. | Day 1, 8 and 15 and day 29/ at count recovery at the end of course 1 (whichever is earlier)
  Mer expression (total and phosphorylated Mer) will be determined using traditional western blotting and/or phospho-flow cytometry in bone marrow and peripheral blood. Mean levels of Mer expression will be calculated at each time point and compared with response at the end of course 1 using repeated measures ANOVA.
Determine the response rate | Day 1-29; qualifying marrow and peripheral counts will be performed within 1 week of each other.
  The response rate is defined by the ability to achieve complete remission (CR) after 1 and 2 courses of this therapy in children with bone marrow relapse of T-ALL or relapsed T-LLy.
Mean time from start of study treatment to transplant in patients with bone marrow relapse of T-ALL or relapsed T-LLy. | Day 1-29
  Time from start of study treatment to transplant in patients with bone marrow relapse of T-ALL or relapsed T-LLy will be recorded, and mean time will be calculated.

CONTACTS AND LOCATIONS:
Overall Officials: Himalee Sabnis, MD, Principal Investigator — Emory University
Locations (4):
- United States (4):
  - Children's Healthcare of Atlanta, Atlanta, Georgia
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Cincinnati Children's Hospital, Cincinnati, Ohio
  - Texas Children's Hospital, Houston, Texas

IPD SHARING:
Plan to Share IPD: Yes
Data related to patient diagnosis, toxicity and outcomes will be shared. Data will be available immediately following publication and will be shared with investigators who propose using the data after being approved by a review committee. Data will be available for the purpose of inclusion in meta-analysis by contacting the principal investigator at hsabnis@emory.edu, following which a data use agreement will be needed for sharing data.
Supporting Information: Study Protocol
Time Frame: Data will be available immediately following publication.
Access Criteria: By contacting the principal investigator at hsabnis@emory.edu, following which a data use agreement will be needed for sharing data.